CLINICAL TRIAL: NCT00568568
Title: Metabolic Studies- Interactions Between GH and Insulin in GHDA. Insulin Resistance and GH Treatment: Dependence of Ambient GH Level Among Patients Treated With GH and Healthy Control Subjects
Brief Title: Metabolic Studies- Interactions Between GH and Insulin in GHDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: M-20070176
Record Dates: First submitted 2007-12-05; First posted 2007-12-06 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Insulin Resistance
Keywords: Growth Hormone; GH signaling; Insulin resistance; Insulin Signaling
MeSH Terms: conditions — Insulin Resistance | interventions — Growth Hormone; Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Growth hormone (Experimental)
  Interventions: Drug: Growth hormone

INTERVENTIONS:
Drug: Growth hormone — GH infusion from 8.00 pm to 03.00 am (dose 10,2 ng/kg/min) c) GH infusion from 02.00 am to 09.00 am (dose 10,2 ng/kg/min).
  Other Names: Norditropin, Novo Nordisk

SUMMARY:
The purpose og this study is to investigate the effects of growth hormon on insulin signalling pathways and the temporal association between administration of GH and developing of insulin resistance.

DETAILED DESCRIPTION:
Insulin resistance is a pathophysiological component of type 2 diabetes, obesity and elevated blood pressure. Overall they are syndromes with multifactorial ethology and partly unclarified pathophysiology. Insulin resistance also occur in more seldom diseases with a more unified pathogenesis. Growth hormone deficiency (GHD) in adults with hypopituitarism is an example of one of those seldom diseases. Prolonged GHD is associated with abdominal overweight, dyslipidemia and increased cardiovascular morbidity. Besides, GHD-patients have decreased insulin sensitivity presumably secondary to the altered body composition. Long term effects of GH-substitution improves insulin sensitivity but it is well-known that subcutaneous administration of GH acute worsen insulin sensitivity in both muscles- and liver-tissue. Recently it has been reported that insulin resistance in patients with type 2 diabetes is associated with the induction of a signal protein called suppressor of cytokine signalling (SOCS). It´s interesting that GH also induces a stimulation of SOCS.

ELIGIBILITY:
Inclusion Criteria:

* Written consent before study start
* Growth Hormone substitution in stable dosis for at least 3 months prior to study start
* Other substitution in stable dosis for at least 3 months prior to study start

Exclusion Criteria:

* Medical treatment for diabetes
* Hypertension even with medical treatment
* BMI > 30
* Excessive alcohol abuse

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-12; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Socs 1-3 activity in muscle tissue and degree of insulin resistance | 6 hours

SECONDARY OUTCOMES:
Growth Hormone Signaling Proteins in Muscle Tissue and other Insulin Signaling Proteins in Muscle Tissue | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jens Otto L Jørgensen, MD, DMSc, Principal Investigator — Depatment M (endocrinology and diabetes), Aarhus University Hospital, Nørrebrogade 44, 8000 Aarhus C, Denmark
Locations (1):
- Department M (endocrinology and diabets), Aarhus, Aarhus, Denmark